CLINICAL TRIAL: NCT00253747
Title: A Pilot Study of Osmotic-Release Methylphenidate in Initiating and Maintaining Abstinence in Smokers With ADHD
Brief Title: Smoking Cessation for Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Eugene Somoza, Adjunct Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-CTN-0029; 5U10DA013732 (NIH)
Record Dates: First submitted 2005-11-13; First posted 2005-11-15 (Estimated); Results first posted 2012-09-17 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-08

CONDITIONS: ADHD; Smoking
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Smoking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Osmotic-Release Methylphenidate (Active Comparator)
  Interventions: Drug: Osmotic-Release Methylphenidate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Osmotic-Release Methylphenidate — OROS-MPH dosing strategy will start with 18 mg/day for 3 days, increasing to 36mg/day for the next three days; increasing to 54 mg/day in week two, and to 72 mg/day in week three through the remainder of the study (as tolerated). And, nicotine patch dosing schedule will be 21 mg/day during weeks 4-11; 14 mg/day during weeks 12-13; and 7 mg/day in week 14.
  Arms: Osmotic-Release Methylphenidate
Drug: Placebo — OROS-MPH (placebo) dosing strategy will start with 18 mg/day for 3 days, increasing to 36mg/day for the next three days; increasing to 54 mg/day in week two, and to 72 mg/day in week three through the remainder of the study (as tolerated). And, nicotine patch dosing schedule will be 21 mg/day during weeks 4-11; 14 mg/day during weeks 12-13; and 7 mg/day in week 14.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate whether Osmotic-Release Methylphenidate (OROS MPH), relative to placebo, increases the effectiveness of standard smoking treatment (i.e., nicotine patch and individual smoking cessation counseling) in obtaining prolonged abstinence for smokers with Attention Deficit Hyperactivity Disorder (ADHD).

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate whether OROS MPH (Concerta), relative to placebo, increases the effectiveness of standard smoking treatment (i.e., nicotine patch and individual smoking cessation counseling) in obtaining prolonged abstinence for smokers with ADHD. The study will involve an estimated 252 participants, recruited from approximately 6 sites.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ADHD2
* Smoked cigarettes for at least 3 months
* Currently smoking > 10 cigarettes/day
* Have an interest in quitting
* Negative urine screen for cocaine, methamphetamine, opiates, benzodiazepines, and marijuana

Exclusion Criteria:

* Have a clinical diagnosis for current abuse or dependence for any psychoactive substance other than nicotine, depression, or anxiety; or a life-time clinical diagnosis of psychosis or bipolar disorder
* Allergic to OROS-MPH
* Pregnant or breastfeeding
* Abnormal electrocardiogram (ECG)
* Taking a Monoamine Oxidase (MAO) Inhibitor
* Taking any medication used for treating either ADHD or smoking
* Use of tobacco products other than cigarettes in the past week
* Blood pressure readings greater than 135/85 and/or a heart rate more than 90 beats per minute on three consecutive clinic visits

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 255 (Actual)
Dates: Start 2005-11; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Somoza, M.D., Ph.D., Principal Investigator — University of Cincinnati; Theresa Winhusen, Ph.D., Principal Investigator — University of Cincinnati
Locations (6):
- United States (6):
  - Massachusetts General Hospital, Cambridge, Massachusetts
  - Mayo Clinic Nicotine Research Program, Rochester, Minnesota
  - VA New York Harbor Healthcare System, New York, New York
  - New York State Psychiatric Institute - Smoking Cessation Program, New York, New York
  - Maryhaven, Inc., Columbus, Ohio
  - Kaiser Permanente (Center for Health Research), Portland, Oregon

REFERENCES:
- [Derived] Luo SX, Wall M, Covey L, Hu MC, Scodes JM, Levin FR, Nunes EV, Winhusen T. Exploring longitudinal course and treatment-baseline severity interactions in secondary outcomes of smoking cessation treatment in individuals with attention-deficit hyperactivity disorder. Am J Drug Alcohol Abuse. 2018;44(6):653-659. doi: 10.1080/00952990.2017.1416474. Epub 2018 Jan 25. PMID 29370538
- [Derived] Covey LS, Hu MC, Winhusen T, Lima J, Berlin I, Nunes E. Anxiety and Depressed Mood Decline Following Smoking Abstinence in Adult Smokers with Attention Deficit Hyperactivity Disorder. J Subst Abuse Treat. 2015 Dec;59:104-8. doi: 10.1016/j.jsat.2015.07.004. Epub 2015 Jul 17. PMID 26272693
- [Derived] Luo SX, Covey LS, Hu MC, Levin FR, Nunes EV, Winhusen TM. Toward personalized smoking-cessation treatment: Using a predictive modeling approach to guide decisions regarding stimulant medication treatment of attention-deficit/hyperactivity disorder (ADHD) in smokers. Am J Addict. 2015 Jun;24(4):348-56. doi: 10.1111/ajad.12193. Epub 2015 Feb 6. PMID 25659348
- [Derived] Nunes EV, Covey LS, Brigham G, Hu MC, Levin FR, Somoza EC, Winhusen TM. Treating nicotine dependence by targeting attention-deficit/ hyperactivity disorder (ADHD) with OROS methylphenidate: the role of baseline ADHD severity and treatment response. J Clin Psychiatry. 2013 Oct;74(10):983-90. doi: 10.4088/JCP.12m08155. PMID 24229749
- [Derived] Westover AN, Nakonezny PA, Winhusen T, Adinoff B, Vongpatanasin W. Risk of methylphenidate-induced prehypertension in normotensive adult smokers with attention deficit hyperactivity disorder. J Clin Hypertens (Greenwich). 2013 Feb;15(2):124-32. doi: 10.1111/jch.12039. Epub 2012 Dec 14. PMID 23339731
- [Derived] Heffner JL, Lewis DF, Winhusen TM. Osmotic release oral system methylphenidate prevents weight gain during a smoking-cessation attempt in adults with ADHD. Nicotine Tob Res. 2013 Feb;15(2):583-7. doi: 10.1093/ntr/nts152. Epub 2012 Sep 6. PMID 22955246
- [Derived] Winhusen TM, Somoza EC, Brigham GS, Liu DS, Green CA, Covey LS, Croghan IT, Adler LA, Weiss RD, Leimberger JD, Lewis DF, Dorer EM. Impact of attention-deficit/hyperactivity disorder (ADHD) treatment on smoking cessation intervention in ADHD smokers: a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2010 Dec;71(12):1680-8. doi: 10.4088/JCP.09m05089gry. Epub 2010 May 18. PMID 20492837
- [Derived] Covey LS, Hu MC, Winhusen T, Weissman J, Berlin I, Nunes EV. OROS-methylphenidate or placebo for adult smokers with attention deficit hyperactivity disorder: racial/ethnic differences. Drug Alcohol Depend. 2010 Jul 1;110(1-2):156-9. doi: 10.1016/j.drugalcdep.2010.02.002. Epub 2010 Mar 12. PMID 20219292

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted by the National Institute on Drug Abuse (NIDA) Clinical Trials Network (CTN) between December 2005 and January 2008. Six study sites recruited participants: 2 substance abuse community treatment programs, 2 Attention Deficit Hyperactivity Disorder (ADHD) clinics and 2 smoking cessation clinics.
Groups:
- Osmotic-Release Methylphenidate (OROS-MPH): For OROS-MPH, the starting dose of 18 mg/day was escalated during the first two study weeks to a maximum of 72 mg/day or to the highest dose tolerated. A trained interventionist provided each participant with a weekly 10 minute smoking cessation counseling session during study weeks 1-11. All participants received transdermal nicotine patches.
- Osmotic-Release Methylphenidate (OROS-MPH) - Placebo: OROS-MPH/placebo was taken through the week 11 visit. A trained interventionist provided each participant with a weekly 10 minute smoking cessation counseling session during study weeks 1-11. All participants received transdermal nicotine patches.
Period: Overall Study
Arm/Group | Osmotic-Release Methylphenidate (OROS-MPH) | Osmotic-Release Methylphenidate (OROS-MPH) - Placebo
Started | 127 | 128
Completed | 103 | 101
Not Completed | 24 | 27
Not completed — Lost to Follow-up | 13 | 14
Not completed — Withdrawal by Subject | 10 | 11
Not completed — Administrative Discharge (1), Other (2) | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Osmotic-Release Methylphenidate (OROS-MPH) | Osmotic-Release Methylphenidate (OROS-MPH) - Placebo | Total
Number analyzed (Participants) | 127 | 128 | 255
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 127 | 128 | 255
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.1 (10.4) | 37.5 (9.6) | 37.8 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 61 | 111
  Male | 77 | 67 | 144
Region of Enrollment [Number; unit: participants]
  United States | 127 | 128 | 255

OUTCOME MEASURES:

1. Primary Outcome: Prolonged Abstinence
Description: The smoking quit date was considered the first day of the O-MPH/P-Stnd Smoking Tx phase, which lasted for 6 weeks or more precisely 42 days (i.e., approximately weeks 5-10). The grace period was the first two weeks (i.e., days 1-14) with the remaining four weeks (days 15-42) comprising the period in which the participant must not meet criteria for treatment failure in order to be scored as obtaining prolonged abstinence. Self-report of cigarette use was assessed using a time-line follow-back (TLFB) assessment using carbon monoxide (CO)levels to correct self-reported smoking days. "Smoking days" were determined by starting with self-reported smoking and non-smoking days and using CO levels measured at weekly visits to modify the self-reports.
Time Frame: Weeks 7-10
Population: Randomized participants who complete at least two visits during the first four weeks following randomization, who reach the full dose of OROS-MPH /Placebo, who have a OROS-MPH /placebo medication compliance rate of at least 75% each week for study weeks 4 through 10, and who attend at least one meeting after initiating the nicotine patch.
Measure: Number; unit: participants
Arm/Group | Osmotic-Release Methylphenidate (OROS-MPH) | Osmotic-Release Methylphenidate (OROS-MPH) - Placebo
Number analyzed (Participants) | 38 | 42
participants | 25 | 28

2. Secondary Outcome: Diagnostic and Statistical Manual-IV(DSM-IV) ADHD Rating Scale
Description: A Generalized Estimating Equations(GEE)model which included treatment group, week, site, and treatment by week and site by week interaction effects was used to compare the groups on the DSM-IV ADHD total severity score (18 domains score at severity levels of 0[none]-3[severe]; maximum score 54) as measured at screening/baseline and study weeks 1-4 using the the interviewer-administered DSM-IV checklist and by the severity portion of the National Institute of Mental Health Clinical Global Impression (CGI) scale to rate the severity of the participant's ADHD symptoms. A single severity score ranging from 1 to 7 is yielded by the CGI severity scale.
Time Frame: Baseline and Study weeks 1,4,7,9,11
Population: Evaluable participants determined using criteria for same in the primary outcome.
Measure: Mean (Standard Deviation); unit: DSM IV ADHD Score
Groups:
- Osmotic-Release Methylphenidate (OROS-MPH)-Baseline; Osmotic-Release Methylphenidate (OROS-MPH)-Week 11; Release Methylphenidate (OROS-MPH)-Week 4; Release Methylphenidate (OROS-MPH)-Week 7: For OROS-MPH, the starting dose of 18 mg/day was escalated during the first two study weeks to a maximum of 72 mg/day or to the highest dose tolerated. A trained interventionist provided each participant with a weekly 10 minute smoking cessation counseling session during study weeks 1-11. All participants received transdermal nicotine patches.
- Osmotic-Release Methylphenidate (OROS-MPH) - Placebo-Baseline; Osmotic-Release Methylphenidate (OROS-MPH) - Placebo-Week 11; Osmotic-Release Methylphenidate (OROS-MPH) - Placebo-Week 4; Osmotic-Release Methylphenidate (OROS-MPH) - Placebo-Week 7; Methylphenidate (OROS-MPH) - Placebo-Week 9: OROS-MPH/placebo was taken through the week 11 visit. A trained interventionist provided each participant with a weekly 10 minute smoking cessation counseling session during study weeks 1-11. All participants received transdermal nicotine patches.
- Release Methylphenidate (OROS-MPH)-Week 9: OROS-MPH, the starting dose of 18 mg/day was escalated during the first two study weeks to a maximum of 72 mg/day or to the highest dose tolerated. A trained interventionist provided each participant with a weekly 10 minute smoking cessation counseling session during study weeks 1-11. All participants received transdermal nicotine patches.
Arm/Group | Osmotic-Release Methylphenidate (OROS-MPH)-Baseline | Osmotic-Release Methylphenidate (OROS-MPH) - Placebo-Baseline | Osmotic-Release Methylphenidate (OROS-MPH)-Week 11 | Osmotic-Release Methylphenidate (OROS-MPH) - Placebo-Week 11 | Release Methylphenidate (OROS-MPH)-Week 4 | Osmotic-Release Methylphenidate (OROS-MPH) - Placebo-Week 4 | Release Methylphenidate (OROS-MPH)-Week 7 | Osmotic-Release Methylphenidate (OROS-MPH) - Placebo-Week 7 | Release Methylphenidate (OROS-MPH)-Week 9 | Methylphenidate (OROS-MPH) - Placebo-Week 9
Number analyzed (Participants) | 38 | 42 | 38 | 42 | 37 | 42 | 35 | 42 | 36 | 40
DSM IV ADHD Score | 38.4 (7.6) | 36.6 (7.7) | 16.4 (12.2) | 24.2 (23.0) | 20.4 (12.6) | 27.2 (12.0) | 20 (12.6) | 24 (13.3) | 17.3 (12.6) | 23.9 (13.6)

3. Secondary Outcome: Point-prevalence Abstinence
Description: A logistic regression including site and treatment group will be used to model rates of achieving point prevalence abstinence as assessed at the final visit of the O-MPH/P-Stnd Smoking Tx phase. Point prevalence abstinence was defined as not smoking in the previous seven days based on self-report using the TLFB method and confirmed with a Carbon Monoxide (CO) level <8 ppm.
Time Frame: Week 11
Population: Evaluable population determined as for primary outcome.
Measure: Number; unit: participants
Arm/Group | Osmotic-Release Methylphenidate (OROS-MPH) | Osmotic-Release Methylphenidate (OROS-MPH) - Placebo
Number analyzed (Participants) | 38 | 42
participants | 24 | 26

ADVERSE EVENTS:
Arm/Group | Osmotic-Release Methylphenidate (OROS-MPH) | Osmotic-Release Methylphenidate (OROS-MPH) - Placebo
Serious Adverse Events (participants affected / at risk) | 2/127 | 0/128
Other Adverse Events (participants affected / at risk) | 35/127 | 28/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osmotic-Release Methylphenidate (OROS-MPH) (N=127) | Osmotic-Release Methylphenidate (OROS-MPH) - Placebo (N=128)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Hospitalized following car accident, not related, study agent temporarily discontinued
Depression (Psychiatric disorders) | 1 (1) | 0 (0) — Hospitalized for worsening of pre-existing depression, not related, no action taken regarding study agent.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osmotic-Release Methylphenidate (OROS-MPH) (N=127) | Osmotic-Release Methylphenidate (OROS-MPH) - Placebo (N=128)
Headache (Nervous system disorders) | 35 (35) | 28 (28)
Nervousness (Psychiatric disorders) | 28 (28) | 21 (21)
Anxiety (Psychiatric disorders) | 24 (24) | 18 (18)
Insomnia (Psychiatric disorders) | 22 (22) | 17 (17)
Nasopharyngitis (Infections and infestations) | 20 (20) | 14 (14)
Decreased Appetite (Metabolism and nutrition disorders) | 23 (23) | 7 (7)
Nausea (Gastrointestinal disorders) | 18 (18) | 10 (10)
Dry Mouth (Gastrointestinal disorders) | 15 (15) | 7 (7)
Abnormal Dreams (Psychiatric disorders) | 9 (9) | 9 (9)
Upper Respiratory Tract Infection (Infections and infestations) | 7 (7) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 10 (10) | 4 (4)
Initial Insomnia (Psychiatric disorders) | 9 (9) | 5 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (6)
Dizziness (Nervous system disorders) | 8 (8) | 5 (5)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7)
Toothache (Gastrointestinal disorders) | 5 (5) | 6 (6)
Stress (Psychiatric disorders) | 5 (5) | 6 (6)
Agitation (Psychiatric disorders) | 5 (5) | 5 (5)
Sleep Disorder (Psychiatric disorders) | 5 (5) | 5 (5)
Psychomotor Hyperactivity (Nervous system disorders) | 9 (9) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 9 (9) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6)
Heart Rate Increased (Investigations) | 9 (9) | 1 (1)
Palpitations (Cardiac disorders) | 9 (9) | 1 (1)
Depressed Mood (Psychiatric disorders) | 3 (3) | 6 (6)
Application Site Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
Dysgeusia (General disorders) | 4 (4) | 4 (4)
Vomiting (Gastrointestinal disorders) | 6 (6) | 2 (2)
Arthalagia (General disorders) | 4 (4) | 4 (4)
Fatigue (General disorders) | 15 (15) | 12 (12)
Depression (Psychiatric disorders) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No